CLINICAL TRIAL: NCT01594801
Title: Testing the Effect of the InsuPad Device in Daily Life Conditions - The InsuPad in Daily Life Study
Brief Title: Testing the Effect of the InsuPad Device in Daily Life Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insuline Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-PP-003
Record Dates: First submitted 2012-05-06; First posted 2012-05-09 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Diabetics Mellitus Type 1; Diabetes Mellitus Type 2
Keywords: DM; insulin; injections
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Subject continue their routine therapy
- Test (Experimental): Subjects using the InsuPad device
  Interventions: Device: InsuPad

INTERVENTIONS:
Device: InsuPad — Use of the InsuPad for at least 3 times a day.
  Arms: Test

SUMMARY:
This is the test protocol for the InsuPad device. The aim of the study is to show economical benefit when using the InsuPad device, by testing the effect of the InsuPad device on reducing injected insulin dose while keeping the same overall glycaemic control.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 to 75 years (including 18 and 75 years old).
* Type 1 or type 2 diabetes mellitus subjects with daily short-acting prandial insulin intake of > 60 IU/day.
* HbA1c >=6.0% and =< 8%
* Use of short-acting prandial insulin analogues with multiple daily injections. The analog insulin brands to be used will be either insulin Lispro (Humalog, Liprolog) or insulin Aspart (NovoRapid) or insulin Glulisin (Apidra).
* Subject agrees to sign consent form before any study-specific tests or procedures are to be performed.
* Study subject is willing to perform at least 5 blood glucose measurements per day for at least 3 months, willing to comply with study procedures and to keep a detailed patient log book.

Exclusion Criteria:

* Excessive fibrosis, lipo-hypertrophy or eczema at injection sites.
* Known gastro- or enteroparesis.
* Unstable chronic disease other than diabetes mellitus (e. g. unstable angina pectoris, renal disease) for the last six months before study start.
* Severe hypoglycaemic events requiring glucagon injection or glucose infusion within the last four weeks prior to study start.
* Hypoglycaemia unawareness (Score > 4 in the Hypoglycaemia Awareness Questionnaire)
* Diabetic ketoacidosis (severe, with hospitalization) within the last six months prior to study start
* Any known life-threatening disease
* Pregnant women, lactating women or women who intend to become pregnant during the observation period
* Any other condition or compliance issues that might interfere with study participation or results
* Subjects with heat sensitivity
* Subjects involved in or planned to participate in other studies
* Subjects who are incapable of contracting or under guardianship

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2012-05; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Efficacy | 3 months
  The primary endpoint of the study is to demonstrate the non-inferiority (margin of 0.4%) for overall glycaemic control defined as HbA1c of a treatment regimen applying InsuPad combined with an insulin dose reduction of >10% in the test group compared to the control group not using InsuPad.
Safety | 3 months
  compare the Frequency of mild hypoglycaemia events (Blood Glucose < 63 mg/dl or 3. 5 mmol/l) with InsuPad and without InsuPad.

CONTACTS AND LOCATIONS:
Locations (9):
- Germany (9):
  - Gemeinschaftspraxis Dr. Klausmann/ Dr. Welslau, Aschaffenburg
  - Diabeteszentrum Bad Mergentheim, Bad Mergentheim
  - ikfe GmbH, Berlin, Berlin
  - GWT-TUD GmbH, Zentrum für Klinische Studien, Dresden
  - ikfe GmbH Mainz, Mainz
  - Zentrum Für Klinische Studien Neuwied, Neuwied
  - ikfe GmbH, Potsdam, Potsdam
  - Dr. Notghi Clinical Trials, Potsdam
  - Allgemeinärztliche Berufsausübungs-gemeinschaft Waldfischbach-Burgalben, Waldfischbach-Burgalben

REFERENCES:
- [Derived] Pfutzner A, Hermanns N, Funke K, Forst T, Behnke T, Bitton G, Nagar R, Raz I, Haak T. The Barmer study: impact of standardized warming of the injection site to enhance insulin absorption and reduce prandial insulin requirements and hypoglycemia in obese patients with diabetes mellitus. Curr Med Res Opin. 2014 May;30(5):753-60. doi: 10.1185/03007995.2014.880049. Epub 2014 Jan 17. PMID 24392996
- See also: Related Info — http://insuline-medical.com